CLINICAL TRIAL: NCT00747526
Title: A Pharmacokinetic, Pharmacodynamic and Safety Study of Single and Multiple Doses of Rabeprazole in Pediatric Subjects With GERD 1 to 11 Months Old, Inclusive
Brief Title: A Study of Single and Multiple Doses of Rabeprazole in Pediatric Patients With Gastroesophageal Reflux Disease (GERD) 1 to 11 Months Old, Inclusive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013948; RABGRD1003 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); 2008-000452-27 (EudraCT Number)
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease (GERD); Pediatrics; Pharmacokinetics; Pharmacodynamics; Rabeprazole; GERD; Aciphex
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rabeprazole sodium 5 mg (Experimental)
  Interventions: Drug: Rabeprazole sodium 5 mg
- Rabeprazole sodium 10 mg (Experimental)
  Interventions: Drug: Rabeprazole sodium 10 mg

INTERVENTIONS:
Drug: Rabeprazole sodium 5 mg — Type= exact number, unit= mg, number= 5, format= bead suspension formulation, route= oral use. Rabeprazole sodium 0.5 mg/kg (using increments of 1 mg dose) once daily from Day 1 to Day 5; possible extension using 5 mg once daily up to 28 consecutive days.
  Arms: Rabeprazole sodium 5 mg
Drug: Rabeprazole sodium 10 mg — Type= exact number, unit= mg, number= 10, format= bead suspension formulation, route= oral use. Rabeprazole sodium 0.5 mg/kg (using increments of 1 mg dose) once daily from Day 1 to up to Day 14; possible extension using 10 mg once daily up to 28 consecutive days.
  Arms: Rabeprazole sodium 10 mg

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (how the drug is absorbed in the body, how it is distributed within the body and removed from the body over time), pharmacodynamics (how the study medication affects the body) and safety of rabeprazole after single and multiple daily administration in infants between the ages of 1 and 11 months, inclusive, with Gastroesophageal Reflux Disease (GERD).

DETAILED DESCRIPTION:
This is an open-label (both physician and patient know the name of the study medication), multicenter, Phase I study, consisting of 2 parts. The first part of the study will be nonrandomized (study drug is intentionally assigned), and all patients will receive the same dose. In the second part of the study, patients will be randomized (study medication assigned by chance) into 2 dose groups. The purpose of the study is to evaluate the pharmacokinetics (PK), pharmacodynamics (intraesophageal/intragastric pH, clinical global impression, formulation palatability and Gastroesophageal Reflux Disease (GERD) daily symptom diary) and safety of rabeprazole after single and multiple daily administration at 2 dose levels in children between the ages of 1 and 11 months, inclusive (up to 11 months 29 days), with GERD. As this study is an exploratory assessment of the PK, pharmacodynamics and safety of rabeprazole in children, no formal hypothesis testing is applied. Safety and tolerability, including monitoring of adverse events, clinical laboratory results, physical examination, vital signs and electrocardiogram measurements (the measuring of the electrical currents in the heart), will be evaluated throughout the study. Patients will receive rabeprazole sodium as single daily oral doses for 5 successive days (Option 1), or up to 14 successive days (10 days minimum) (Option 2) as a bead formulation. In Part 1, patients will receive single and multiple daily (every 24 hours) doses of 0.5 mg/kg, using increments of 1 mg dose. Safety and PK data from Part 1 of the study will determine the 2 dosages to be studied in Part 2 of the study. In Part 2, patients may receive rabeprazole sodium as single daily oral doses for up to a maximum of 28 consecutive days as a bead formulation. Patients will be randomized into either the 5 mg dose or 10 mg dose group.

ELIGIBILITY:
Inclusion Criteria:

* Minimum weight of 5 kg (treatment Option 1) or 3 kg (treatment Option 2) with a diagnosis of GERD
* Informed consent signed by at least one parent
* Patients who have been treated with, or are currently receiving a proton pump inhibitor (PPI), H2 blockers, or antacids are eligible (as long as they can go off antacids for 24 hours, and PPIs and H2 blockers for three days prior to dosing, except for cimetidine, which must be discontinued for at least seven days prior to dosing) and remain off these medications for the treatment period

Exclusion Criteria:

* Patients who have history of or current clinically significant medical illness (excluding GERD) including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, infection, or any other illness that the investigator considers should exclude the patient or that could interfere with the interpretation of the study results
* Primary pulmonary or ears, nose, and throat (ENT) symptoms
* History of or current presence of peptic ulcers
* Presence of "warning signals", suggesting cause of vomiting/regurgitation other than GERD
* Any condition which would make the patient, in the opinion of the Investigator or Sponsor, unsuitable for the study

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2007-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | At Days 1, 5, and 10
Pharmacodynamic parameters | At Days 1, 5, and 10

SECONDARY OUTCOMES:
Number of Patients with Adverse Events as a Measure of Safety | Approximately 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Development, L.L.C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (20):
- United States (13):
  - Little Rock, Arkansas
  - Oakland, California
  - Washington D.C., District of Columbia
  - Maitland, Florida
  - Louisville, Kentucky
  - Jackson, Mississippi
  - Bridgeton, Missouri
  - Long Branch, New Jersey
  - Greenville, North Carolina
  - Cleveland, Ohio
  - Toledo, Ohio
  - Youngstown, Ohio
  - Houston, Texas
- Belgium (2):
  - Antwerp
  - Brussels
- São Paulo, Brazil
- Poland (2):
  - Lublin
  - Warsaw
- United Kingdom (2):
  - Barnsley
  - London

REFERENCES:
- [Derived] Treem W, Hu P, Sloan S. Normal and proton pump inhibitor-mediated gastrin levels in infants 1 to 11 months old. J Pediatr Gastroenterol Nutr. 2013 Oct;57(4):520-6. doi: 10.1097/MPG.0b013e31829b6914. PMID 23689261
- See also: A Pharmacokinetic, Pharmacodynamic, and Safety Study of Single- and Multiple Doses of Rabeprazole in Pediatric Subjects with GERD 1 to 11 Months old, Inclusive — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=765&filename=CR013948_CSR.pdf